CLINICAL TRIAL: NCT06418477
Title: Daratumumab, Bortezomib, Cyclophosphamide, and Dexamethasone Therapy for Patients with Monoclonal Immunoglobulin Deposition Disease
Brief Title: Daratumumab, Bortezomib, Cyclophosphamide, and Dexamethasone Therapy for Patients with MIDD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jin Lu, MD, Principal Investigator, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024PHB134-001
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Monoclonal Gammopathy of Renal Significance
Keywords: Daratumumab; Bortezomib; Monoclonal Immunoglobulin Deposition Disease
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dara-CyBorD (Experimental): Daratumumab:
  Cyclophosphamide Bortezomib Dexamethasone
  Interventions: Drug: Dara-CyBorD

INTERVENTIONS:
Drug: Dara-CyBorD — Patient will receive Dara-CyBorD (Daratumumab, Bortezomib, Cyclophosphamide, Dexamethasone) for at least 6 cycles, and then Daratumumab maintainance.
  Drug: Daratumumab: 16mg/kg IV dose OR 1800 mg subcutaneously Drug: Cyclophosphamide: 300 mg/m^2 as an oral or IV dose Drug: Bortezomib: 1.3 mg/m^2 as an subcutaneous (SC) injection. Drug: Dexamethasone: 20-40mg Patients will receive the above drugs (Dara-CyBorD) on Days 1, 8, 15, 22 in every 28-day cycle for a maximum of 6 cycles. Daratumumab will be administered weekly for the first 8 weeks (2 cycles), then every 2 weeks for 4 cycles (cycles 3-6), and then every 4 weeks until progression of disease or subsequent therapy for a maximum of 1 years.
  Note: If patients achieve less than hematologic VGPR by cycle 3 or less than PR by cycle 2, treatment plan will be allowed to discontinued, according to treatment principle in systemic light chain amyloidosis.

SUMMARY:
This is an open-label, multicenter, Phase 2 study in subjects with newly diagnosed monoclonal immunoglobulin deposition disease treated with daratumumab, bortezomib, cyclophosphamide, and dexamethasone.

DETAILED DESCRIPTION:
The current study aims to investigate daratumumab, bortezomib, cyclophosphamide, and dexamethasone regimen in patients with newly diagnosed monoclonal immunoglobulin deposition disease. Approximately 25 subjects will receive primary therapy with daratumumab-CyBorD. The primary endpoint is overall complete hematologic response (CHR) rate at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of monoclonal immunoglobulin deposition disease without anti-plasma cell treatment
2. ECOG 0,1,2
3. Neu≥ 1.0*10^9/L, HGB ≥70g/L, PLT ≥ 50*10^9/L.
4. Total bilirubin (TBil) ≤3×upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0×ULN;
5. Informed consent explained to, understood by and signed by the patient.

Exclusion Criteria:

1. Prior therapy for MIDD, with the exception of equal or less than 160 mg dexamethasone (or equivalent corticosteroid)
2. Fulfill with the criteria of active multiple myeloma or active lymphoplasmacytic lymphoma.
3. Presence of other tumors which is/are in advanced malignant stage and has/have systemic metastasis;
4. Severe or persistent infection that cannot be effectively controlled;
5. Presence of severe autoimmune diseases or immunodeficiency disease;
6. Patients with active hepatitis B or hepatitis C ([HBVDNA+] or [HCVRNA+]);
7. Patients with HIV infection or syphilis infection;
8. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Hematologic Complete Response at the completion of 6 cycles | 6 months
  Hematologic complete response requires absence of monoclonal protein by immunofixation electrophoreses of both serum and urine as well as a normal FLC ratio (FLCr). CR is considered when FLCr was altered in favour of the non-amyloidogenic, uninvolved FLC (uFLC), even though the ratio may not have been normalised.

SECONDARY OUTCOMES:
Rate of Hematologic CR (Complete Response)+ VGPR (very good partial response) at the completion of 6 cyels | 6 months
Rate of Hematologic ORR (Overall Response, CR+VGPR+low-dFLC response+PR) at the completion of 6 cyels | 6 months
Renal response at 6 months | 6 months
  Renal response at 6 months
Cardiac response at 6 months | 6 months
  Cardiac response (for patients with cardiac involvement) at 6 months
MRD status at 6 months | 6 months
  Minimal residual disease status at 6 months
Renal Survival in 2 years | 2 years
  Renal Survival in 2 years
Overall Survival in 2 years | 2 years
  Overall Survival in 2 years
TRAEs | 2 years
  Treatment-related adverse events up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, Principal Investigator — Peking University People's Hospital
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No